CLINICAL TRIAL: NCT01557686
Title: Patient Activation Through Counseling and Exercise - Acute Leukemia - Pilot Trial
Brief Title: Health Counseling and Exercise in Patients With Acute Leukemia - Pilot Study
Acronym: PACE-AL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitetshospitalernes Center for Sygepleje (Other)
Collaborators: Novo Nordisk A/S (Industry); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Mary Jarden, Research Fellow, Universitetshospitalernes Center for Sygepleje
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-4-2010-046 Pilot
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Acute Leukemia
Keywords: Cancer Related fatigue; Quality of Life; Psychosocial Intervention; Rehabilitation; Physical Fitness; Physical Activity; Exercise Therapy; Exercise; Hematologic; Hematological; Leukemia, Myeloid, Acute; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Acute Leukemia
MeSH Terms: conditions — Motor Activity; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Health counseling and exercise — The intervention is initiated during chemotherapy treatment (consolidation) in the outpatient clinic and continues for 6 weeks. The intervention is a three hour/wk supervised in-hospital programme of aerobic (stationary cycle) and functional muscle training, progressive relaxation training, nutrition supplement (protein and carbohydrate) immediately after training and two health-promoting counseling sessions - Further, patients are fitted with a step counter pedometer.

SUMMARY:
The purpose of this pilot study is to test an exercise-based multidimensional intervention for patients with acute leukaemia undergoing consolidation chemotherapy in the context of outpatient management. Further, to test for safety, feasibility and preliminary effect on physical and functional capacity, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are able to speak Danish > 18 years and newly diagnosed with acute leukæmia (MDS, AML, CMML, APL or ALL)
* Normal EKG, blood pressure and pulse
* Signed informed written consent

Exclusion Criteria:

* Medical reason that contraindicates physical activity
* Patients diagnosed with a symptomatic cardiac disease within the last three months.
* Documented bone metastasis
* Dementia, psychotic
* Cannot write or read Danish
* Patients unable to carry out baseline tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Feasibility - adherence rates | Adherence to the intervention components from baseline to 6 weeks
  Percentage of intervention participation

SECONDARY OUTCOMES:
Adverse events | baseline to 6 weeks
  Number and type of adverse events
6MWD | Change from baseline in 6MWD at 6 weeks
  Change in distance in meter
Attrition | Withdrawal from the project from baseline to 6 weeks
  Number of patients that withdrew from the project
Timed chair stand | Change from baseline in timed chair stand at 6 weeks
  Change in the number of repetitions
Timed bicep curl | Change from baseline in timed bicep curl at 6 weeks
  Change in number of repetitions
FACT-Anemia | Change from baseline in FACT-An at 6 weeks
  Change in scores for quality of life/function
HADS | Change from baseline in HADS at 6 weeks
  Change in scores for emotional wellbeing
SF36 | Change from baseline in SF36 at 6 weeks
  Change in scores for general health
MDSAI | Change from baseline over time (1,2,3,4,5,6 weeks)
  Change in scores for symptom burden

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jarden, Ph.D., Principal Investigator — Copenhagen University Hospital at Herlev
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen
  - Herlev Hospital, Herlev